CLINICAL TRIAL: NCT02859298
Title: Feasibility Study and Predictive Value of the Uterine Cervix Polarimetric Imaging for the Management of the Threat of Premature Delivery : The POLARMAP Project
Brief Title: Feasibility Study and Predictive Value of the Uterine Cervix Polarimetric Imaging for the Management of the Threat of Premature Delivery.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of human ressources
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Andre Nazac, Head of clinic, Brugmann University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUB-Polarmap
Record Dates: First submitted 2016-08-04; First posted 2016-08-09 (Estimated); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Premature Delivery
Keywords: Premature Delivery; Polarimetric Imaging; Polarimetric colposcope; Diagnostic tool
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suspicion of threat of premature delivery (Experimental): 10 consecutive patients arriving at the Brugmann maternity with suspicion of a threat of premature delivery will be encouraged to participate in this study, before the onset of any tocolytic treatment. The patient will receive an standard examination of the cervix and at the same time a polarimetric measurement.
  Interventions: Device: Uterine Cervix Polarimetric Imaging
- Normal pregnancy (Active Comparator): 10 control patients, with the same term of pregnancy, will be benefit from the same measurements.
  Interventions: Device: Uterine Cervix Polarimetric Imaging

INTERVENTIONS:
Device: Uterine Cervix Polarimetric Imaging — Polarimetric imaging is a promising optical technique that can provide information in large field and potentially in vivo about the abundance and 3D structure of collagen. Images will be taken with a polarimetric colposcope. As the imaging is realized with visible light from classical sources (lamps or LEDs, neither lasers or other high intensity sources, nor any ionizing UV radiation) and without any chemicals, it is totally innocuous, just like the intensity imaging used in conventional colposcopy.

SUMMARY:
Prematurity is the first cause of perinatal mortality and morbidity worldwide. The threat of premature delivery (TPD), the most important complication and the leading cause of hospitalization during pregnancy has multiple origins which are seldom precisely identified.

The standard medical examination for the detection of patients with TPD is the endovaginal ultrasonographic examination of uterine cervix (echography).

Gynaecologists focus on the use of a new low-cost diagnostic tool based on optical imaging technologies with polarized light. The polarization is the spatio-temporal orientation of a wave's electric field. This light property, invisible with the naked eye, is sensitive to the morphological transformations of a tissue and the orientation of collagen fibers. Such tool would not require an extensive training and should provide an objective quantitative result with a sensitivity and specificity greater than conventional ultrasonography. This would be a considerable contribution to the health care of TPD, a real societal problem in Belgium, Europe and all over the world.

The POLARMAP project proposes the possibility to observe in vivo and during pregnancy, the structural evolution, the density and the orientation changes of collagen fibers. A relevant scoring of collagen status might provide an alternative, and potentially objective and accurate quantifier of the time left before delivery.

DETAILED DESCRIPTION:
Prematurity is the first cause of perinatal mortality and morbidity worldwide. The threat of premature delivery (TPD), the most important complication and the leading cause of hospitalization during pregnancy has multiple origins which are seldom precisely identified.

In Belgium and Europe, the estimated rate of premature births is about 10 %. This rate has been stable over the last two decades in spite of the introduction of new tocolytic treatments and the use of cervical length measurement by transvaginal ultrasound to assess the risk of preterm birth.

The standard medical examination for the detection of patients with TPD is the endovaginal ultrasonographic examination of uterine cervix (echography). Ultrasound examination is more accurate and reproducible compared to cervical digital one, and it possesses two essential qualities of a diagnostic examination: it is easily accepted by the patients and the learning curve is fast.

This technique is validated with well-known criteria, namely, the shortening of the effective length and the opening of the internal orifice of the cervix. The threshold for these two criteria depends on the practitioner's choice: at 30 mm effective length, the sensitivity and negative predictive values are high, but the specificity is poor, while the opposite is true if the threshold is set at 20 mm.

Ultrasound examination for the identification of the patients at risk of premature delivery is a real improvement over cervical digital examination. However, this technique is not ideal, due to the lack of objective criteria for the choice of threshold, because of the imperfect correlation ("noise") between the measured effective length of uterine cervix and the time left before the birth. Moreover, the use of cervical ultrasonography in the strategy of premature delivery screening is not well established.Finally, the transvaginal ultrasound probes are not available in all perinatal centers that would be yet all concerned in case of preterm delivery.

Gynaecologists focus on the use of a new low-cost diagnostic tool based on optical imaging technologies with polarized light. The polarization is the spatio-temporal orientation of a wave's electric field. This light property, invisible with the naked eye, is sensitive to the morphological transformations of a tissue and the orientation of collagen fibers. Such tool would not require an extensive training and should provide an objective quantitative result with a sensitivity and specificity greater than conventional ultrasonography. This would be a considerable contribution to the health care of TPD, a real societal problem in Belgium, Europe and all over the world.

The POLARMAP project proposes the possibility to observe in vivo and during pregnancy, the structural evolution, the density and the orientation changes of collagen fibers.

During the whole pregnancy and until its very end, the cervix is kept closed by abundant and well-organized collagen (the main structural protein in cervical tissue), when the collagen is partly destroyed and/or disorganized before the onset of labor. These changes in collagen structure, which soften the cervix and allow its opening for child birth, have been seen for both premature and full-term births. A relevant scoring of collagen status might thus provide an alternative, and potentially objective and accurate quantifier of the time left before delivery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* normal pregnancy for control group
* threat of premature delivery after 24 weeks of pregnancy for test group

Exclusion Criteria:

- None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08-09 (Actual); Primary Completion 2018-08-24 (Actual); Study Completion 2018-08-24 (Actual)

PRIMARY OUTCOMES:
Signal to noise ratio | 1 second
  Measure of polarimetric imaging feasibility. Signal to noise ratio in a measurement time compatible with in vivo imaging (less than one second)
Reproducibility (%) | 1 second
  Reproducibility of acquired images (expressed in %)
Lickert scale | 10 minutes
  Measure of the acceptability of the patient (psychometric scale to be filled by the patient)

SECONDARY OUTCOMES:
Retardance | 1 second
  Correlation between retardance (polarimetric parameter) and premature delivery.
Depolarization | 1 second
  Correlation between depolarization (polarimetric parameter) and premature delivery.

CONTACTS AND LOCATIONS:
Overall Officials: André Nazac, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

REFERENCES:
- [Background] Pierangelo A, Nazac A, Benali A, Validire P, Cohen H, Novikova T, Ibrahim BH, Manhas S, Fallet C, Antonelli MR, Martino AD. Polarimetric imaging of uterine cervix: a case study. Opt Express. 2013 Jun 17;21(12):14120-30. doi: 10.1364/OE.21.014120. PMID 23787602
- [Background] Rehbinder J, Haddad H, Deby S, Teig B, Nazac A, Novikova T, Pierangelo A, Moreau F. Ex vivo Mueller polarimetric imaging of the uterine cervix: a first statistical evaluation. J Biomed Opt. 2016 Jul 1;21(7):71113. doi: 10.1117/1.JBO.21.7.071113. PMID 27108592
- [Background] Bancelin S, Nazac A, Ibrahim BH, Dokladal P, Decenciere E, Teig B, Haddad H, Fernandez H, Schanne-Klein MC, De Martino A. Determination of collagen fiber orientation in histological slides using Mueller microscopy and validation by second harmonic generation imaging. Opt Express. 2014 Sep 22;22(19):22561-74. doi: 10.1364/OE.22.022561. PMID 25321725